CLINICAL TRIAL: NCT03837080
Title: Efficacy of Nutrition Education Tailored for Chronic Pain Patients on Pain Intensity and Quality of Life - A Randomized Clinical Trial
Brief Title: Nutrition Intervention for Chronic Pain Patients
Acronym: NutChROPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Ines Banjari, PhD, Associate Prof., Head of Department of Food and Nutrition Research, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JJStrossmayerU
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; nutrition education; inflammatory biomarkers
MeSH Terms: conditions — Chronic Pain | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Cluster randomization (groups of patients will be randomly assigned to the Intervention or the Control arm)
Masking Description: The whole group will be randomized (cluster randomization) to either Intervention or Control arm. Each group consists of 8 to 12 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education (Experimental): Participants suffering from chronic pain enrolled in the 4-week Pain Management Clinic organized at the Department of Anesthesiology, Resuscitation and Intensive Care will go through a series of individual and group nutrition educations. Educations are specifically tailored for chronic pain patients, based on our preliminary findings on this group of patients.
  Interventions: Other: Nutrition Education
- Control (No Intervention): Participants suffering from chronic pain enrolled in the 4-week Pain Management Clinic organized at the Department of Anesthesiology, Resuscitation and Intensive Care. Patients will receive all treatments (e.g. physical therapy) except the nutrition education.

INTERVENTIONS:
Other: Nutrition Education — Every patient will receive one individual and two group counselings on specific nutrition-related recommendations for chronic pain patients.
  Other Names: Chronic Pain Nutrition Education
  Arms: Nutrition Education

SUMMARY:
The primary objective of the study is to determine the effectiveness of nutrition education (individual and group) on the intensity of pain in patients suffering from chronic pain. The secondary goal is to determine whether there is a change in the status of the patient's nutrition, their quality of life, quality of life, and other indicators of the psychophysical condition of the patient.

DETAILED DESCRIPTION:
The underlying hypothesis of the study is that patients with chronic pain that go through a series of nutrition education (individual and group) specifically tailored to fit their needs (based on our preliminary findings), they increase the consumption of foods that have antiinflammatory properties, which will result in lower levels of inflammatory cytokines in the body (high sensitivity C-reactive protein (hs-CRP ), interleukin (IL) -2, IL-4 and IL-6), and consequently reduce the intensity of pain. Also, weight loss in obese patients is expected, and it will have an contributing effect of the intervention. Patient's quality of life and indicators of their psychophysical condition (eg, depression level) are also expected to improve.

Chronic pain patients who either attend Daily clinic (Control Arm) or the 4-week multidisciplinary programme at the Department of Anesthesiology, Resuscitation and Intensive Care (Intervention Arm) will be recruited. They will be followed for total of 8 weeks (4 week intervention + 4 week follow-up).

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* chronic low back pain with or without radiculopathy patients; non-cancer pain
* BMI within the range >18 and <35 kg/m2
* Croatian-speaking
* referred to a multidisciplinary pain management center
* able to report on their health and pain status (neurologically stable)
* pain intensity on 0-10 visual analog scale ≥ 5 prior to treatment
* magnetic resonance imaging (MRI) of the lumbar spine and electromyography (EMNG) studies completed confirming clinical symptoms of low back pain with or without radiculopathy

Exclusion Criteria:

* younger than 18 or older than 80
* cancer pain
* pregnancy
* disability (unable to walk)
* inability to fill in questionnaires in Croatian
* cognitive impairment
* significant, symptomatic uncontrolled psychosis
* psychiatric disorder
* pain intensity on 0-10 visual analog scale < 5 prior to treatment
* severe somatic disorder (oncological disease, type 1 diabetes, hepatological or nephrological)
* undergoing current treatment for a major medical illness such as malignancy, autoimmune or immune deficiency disorder
* acute low back pain, or shorter than 6 months
* clotting disorders
* BMI <18 or over 35 kg/m2
* nutritional deficiency (e.g. iron deficiency anaemia, osteoporosis)
* current or history of eating disorder (anorexia, bulimia or EDNOS)
* current use of weight loss interventions (drugs; exercise interventions)
* regular use of supplemental omega-3 fatty acids, gamma-linolenic acid or vitamin D

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  We will use simple, patient-based pain screening questionnaire called the painDETECT questionnaire (validated and widely used to assess pain intensity in chronic pain patients). The questionnaire is based on the scale from 1 (no pain) to 10 (extreme pain).

SECONDARY OUTCOMES:
Change in high-sensitive C-reactive protein after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  high sensitive C-reactive protein (hs-CRP) (mg/L),
Change in interleukines after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  IL-2 (pg/mL), IL-4 8pg/mL), IL-6 (pg/mL)
Change in monocyte chemoattractant protein after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  Monocyte chemoattractant protein (MCP-1) (pg/mL)

OTHER OUTCOMES:
Change in psychological status after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  Depression, Anxiety and Stress Scale (DASS-21) Questionnaire is a validate questionnaire freely accessible and will be scored according to the instruction manual.
Change in Health-Related Quality of Life after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. Total of 36 questions (items) are scored on a 0 to 100 range where higher score corresponds to better quality of life. Items are divided into a total of 8 scales and assess the following: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain and general health. For each scale scoring is done on a 0 to 100 range where higher scores correspond to better health.
Physical activity and sleep monitoring throughout the intervention and follow-up period | Throughout the intervention and 4 weeks post-intervention
  Wearable Health (fitness) device (MiFit) will be used to track patient's physical activity and sleep duration.
Change in Pain Catastrophizing after the intervention and after 4-week follow-up | At inclusion, 4 weeks after the intervention, 4 weeks post-intervention
  The Pain Catastrophizing Scale (PCS) will be used to determine the change in patient's catastrophizing scale related to pain. The questionnaire is based on a scale from 1 (not at all) to 4 (all the time) and assess patient's preoccupation with the pain. The questionnaire will be scored according to the instruction manual.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Banjari, PhD, Principal Investigator — Department of Food and Nutrition Research, Faculty of Food Technology
Locations (1):
- Department of Food and Nutrition Research, Faculty of Food Technology, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
This project is the doctorate thesis project so all data sharing requests can be submitted after the defense by contacting the PI directly.